CLINICAL TRIAL: NCT00710411
Title: Inflammatory Response in Polytraumatized Patients
Brief Title: Inflammatory Response After Muscle and Skeleton Trauma
Acronym: IRAMST
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, MBA, University of Ulm
Other Study IDs: DFG KFO-200
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Trauma
Keywords: humans; patients; polytrauma; complement; inflammation; inflammatory response; biomarkers; cytokines; cell surface markers; apoptosis; NF-kappaB; functional polymorphisms; mesenchymal stem cell; severity of injury; ISS; infections; systemic inflammatory response syndrome; SIRS; sepsis; severe sepsis; shock; organ dysfunctions; SOFA; severity of disease; APACHEII; SAPSII; SPAPS3; length of stay; wound healing; outcome; mortality
MeSH Terms: conditions — Multiple Trauma; Inflammation; Infections; Systemic Inflammatory Response Syndrome; Sepsis; Shock

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, and tissues will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A, 2: Polytraumatized patients with ISS > 18 and healthy controls

SUMMARY:
The purpose of this study is to determine the inflammatory response after multiple trauma in humans.

DETAILED DESCRIPTION:
Polytraumatized patients are via a systemic inflammatory response syndrome at high risk for an uneventful outcome in the posttraumatic phase. One of the main functions of the inflammatory response is the recognition and elimination of damaged tissues and microorganisms. In polytraumatized patients, a huge amount of damaged cells occurs which has to be eliminated by programmed cell death (apoptosis)without damaging surrounding tissues. It remains unclear whether, when and how an interplay of complement system, NF-kB, danger and pattern recognition receptors, apoptosis, mesenchymal stem cells and their regulation may be beneficial and harmful. Differing activation of the complement system, pro-inflammatory biomarkers and predisposing polymorphisms of response and receptor genes are expected to lead to varying outcome. Therefore, this prospective observational study will enroll n=60 polytraumatized patients with an ISS>18 to monitor longitudinally their inflammatory response after trauma and to find out whether there is a discriminating pattern of the cross talk between complement system, biomarkers and apoptosis in patients with beneficial or harmful outcome.

ELIGIBILITY:
Inclusion Criteria:

* multiple trauma injury, injury severity score (ISS) > 18 with

  1. isolated fractures of the extremities
  2. fractures of the extremities combined with blunt/penetrating visceral trauma
  3. fractures of the extremities combined with blunt/penetrating thoracic trauma
  4. isolated head injury with morphological changes in CCT
  5. combination of points 1 - 4

     Exclusion Criteria:
* life expectancy < 24 hours
* participation in other trials
* ISS < 18
* cardiopulmonary reanimation on the accident scene or dying immediately after hospital admission
* age < 18 years
* known or suspected pregnancy
* patients with ray-treatment or chemotherapy within the last three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Polytraumatized patients with an ISS > 18 Controls: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory pattern of complement activation, biomarkers and complement-regulating proteins (CRegs)on leukocytes | 0, 1, 4, 12, 24, 48, 96, 120 und 240 h after trauma

SECONDARY OUTCOMES:
inflammatory biomarkers, cell surface markers, apoptosis, functional polymorphisms, mesenchymal stem cells, severity of injury (ISS), infections, SIRS, sepsis, shock, organ dysfunctions, severity of disease, ICU length of stay, wound healing, mortality | 0, 1, 4, 12, 24, 48, 96, 120 und 240 h after trauma for biochemical and immunological parameters; ISS on admission; scores on a daily basis; ICU and hospital death on discharge

CONTACTS AND LOCATIONS:
Overall Officials: Manfred M Weiss, MD, MBA, Principal Investigator — Clinic of Anesthesiology, University Hospital Medical School, Steinhoevelstrasse 9, 89070 Ulm, Germany
Locations (1):
- Clinic of Anesthesiology and Clinic of Traumatology, Hand-, Plastic-, and Reconstructive Surgery, Ulm, Germany

REFERENCES:
- [Result] Huber-Lang M, Denk S, Fulda S, Erler E, Kalbitz M, Weckbach S, Schneider EM, Weiss M, Kanse SM, Perl M. Cathepsin D is released after severe tissue trauma in vivo and is capable of generating C5a in vitro. Mol Immunol. 2012 Feb;50(1-2):60-5. doi: 10.1016/j.molimm.2011.12.005. Epub 2012 Jan 14. PMID 22244896
- [Result] Unnewehr H, Rittirsch D, Sarma JV, Zetoune F, Flierl MA, Perl M, Denk S, Weiss M, Schneider ME, Monk PN, Neff T, Mihlan M, Barth H, Gebhard F, Ward PA, Huber-Lang M. Changes and regulation of the C5a receptor on neutrophils during septic shock in humans. J Immunol. 2013 Apr 15;190(8):4215-25. doi: 10.4049/jimmunol.1200534. Epub 2013 Mar 11. PMID 23479227
- [Result] Denk S, Wiegner R, Hones FM, Messerer DA, Radermacher P, Weiss M, Kalbitz M, Ehrnthaller C, Braumuller S, McCook O, Gebhard F, Weckbach S, Huber-Lang M. Early Detection of Junctional Adhesion Molecule-1 (JAM-1) in the Circulation after Experimental and Clinical Polytrauma. Mediators Inflamm. 2015;2015:463950. doi: 10.1155/2015/463950. Epub 2015 Oct 18. PMID 26556956
- [Result] Kozarcanin H, Lood C, Munthe-Fog L, Sandholm K, Hamad OA, Bengtsson AA, Skjoedt MO, Huber-Lang M, Garred P, Ekdahl KN, Nilsson B. The lectin complement pathway serine proteases (MASPs) represent a possible crossroad between the coagulation and complement systems in thromboinflammation. J Thromb Haemost. 2016 Mar;14(3):531-45. doi: 10.1111/jth.13208. Epub 2016 Feb 15. PMID 26614707